CLINICAL TRIAL: NCT02909439
Title: Pulmonary Function, Muscle Strength, Time to Extubation and Quality of Recovery in the Post Anesthesia Care Unit After Reversal of Neuromuscular Blockade With Neostigmine or Sugammadex.
Brief Title: Quality of Recovery After Reversal With Neostigmine or Sugammadex.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ramon Abola, Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 917402-3
Record Dates: First submitted 2016-08-31; First posted 2016-09-21 (Estimated); Results first posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Incomplete Reversal of Neuromuscular Block
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neostigmine (Active Comparator): Patients in this arm will receive neostigmine for reversal of neuromuscular blockade. Neostigmine is historically the medication that has been used for this purpose.
  Interventions: Drug: Neostigmine
- Sugammadex (Active Comparator): Patients in this arm will receive sugammadex for reversal of neuromuscular blockade. Sugammadex is a newer, FDA approved, medication for this purpose.
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — Sugammadex will be given for reversal of neuromuscular blockade.
  Other Names: Bridion
  Arms: Sugammadex
Drug: Neostigmine — Neostigmine will be given for reversal of neuromuscular blockade.
  Other Names: Prostigmine
  Arms: Neostigmine

SUMMARY:
This study will compare patient recovery measures after reversal of neuromuscular blockade with neostigmine or sugammadex after surgery. Measures include pulmonary function, muscle strength, time to extubation and quality of recovery in the post anesthesia care unit.

DETAILED DESCRIPTION:
Sugammadex has been shown to have a faster onset and more reliable reversal of neuromuscular blockade when compared to neostigmine as measured by return of Train-of-four (TOF) ratio to >0.9. (Breuckmann, 2015) The investigator's hypothesis is that sugammadex will be associated with improved deep breathing as measured by incentive spirometry in the PACU. The investigators also hypothesize that patients reversed with sugammadex will have shorter times to extubation and better recovery profiles in the PACU as measured by strength, PACU discharge readiness and quality of recovery scores.

Residual neuromuscular blockade after surgery can result in airway compromise, pulmonary complications, and possible need for reintubation and can be a negative experience for patients. Reintubation after surgery is currently a quality measure in NSQIP (National Surgery Quality Improvement Program) A TOF ratio of <0.9 has been identified as a marker of residual neuromuscular blockade in the PACU. (Farhan 2013) Several clinical trials have shown that reversal of neuromuscular blockade with sugammadex results in a faster and more reliable return to TOF ratio of >0.9 when compared to neostigmine. However most of these studies primarily report on TOF ratios. There are scant data on clinical outcomes after reversal with neostigmine versus sugammadex. Incentive spirometry is a clinically meaningful measurement of postoperative pulmonary function, i.e the ability to breath deeply, which minimizes atelectasis and risk of postoperative pneumonia.

The investigators will compare recovery profiles of patients who have received sugammadex or neostigmine for reversal of neuromuscular blockade after surgery. The primary outcome will be incentive spirometry volumes after surgery as a measure of pulmonary function. The secondary measures include hand grip measured using a dynamometer, time to extubation, time to PACU discharge, time to sit independently, and quality of recovery 15 survey scores.

This will be a single-center, prospective, randomized, assessor blinded, controlled trial. Patients will be randomized to either receive sugammadex or neostigmine for the reversal of neuromuscular blockade. The anesthesiologist will be unblinded to the study drug however the assessor in the PACU will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be willing and able to provide written informed consent for the study
* Participant must be greater than or equal to 18 years of age
* Participant must be ASA (American Society of Anesthesiologists) class I, II or III
* Planned use of neuromuscular blocking drugs
* Planned use of endotracheal intubation
* Planned for extubation to occur in the OR

Exclusion Criteria:

* ASA (American Society of Anesthesiologists) Class IV
* Age < 18 years old
* Inability to give oral or written consent
* Known or suspected neuromuscular disorder impairing neuromuscular function
* True allergy to muscle relaxants
* A (family) history of malignant hyperthermia
* A contraindication for neostigmine or sugammadex administration
* Serum creatinine level of greater than 2.0 mg/dL
* Surgery where the patient's arm is not available for neuromuscular monitoring
* A plan to extubate under deep anesthesia
* Pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-11; Primary Completion 2017-11-09 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Abola, MD, Principal Investigator — Stony Brook Medicine, Department of Anesthesiology
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brueckmann B, Sasaki N, Grobara P, Li MK, Woo T, de Bie J, Maktabi M, Lee J, Kwo J, Pino R, Sabouri AS, McGovern F, Staehr-Rye AK, Eikermann M. Effects of sugammadex on incidence of postoperative residual neuromuscular blockade: a randomized, controlled study. Br J Anaesth. 2015 Nov;115(5):743-51. doi: 10.1093/bja/aev104. Epub 2015 May 2. PMID 25935840
- [Background] Farhan H, Moreno-Duarte I, McLean D, Eikermann M. Residual Paralysis: Does it Influence Outcome After Ambulatory Surgery? Curr Anesthesiol Rep. 2014 Dec;4(4):290-302. doi: 10.1007/s40140-014-0073-6. PMID 25530723
- [Derived] Abola RE, Romeiser J, Rizwan S, Lung B, Gupta R, Bennett-Guerrero E. A randomized-controlled trial of sugammadex versus neostigmine: impact on early postoperative strength. Can J Anaesth. 2020 Aug;67(8):959-969. doi: 10.1007/s12630-020-01695-4. Epub 2020 May 13. PMID 32405975

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 patients were excluded after enrollment. The reasons were (1) no longer met inclusion criteria (n =10), declined to participate (n=3), change in surgical date & logistical issues (n=5)
Period: Overall Study
Arm/Group | Neostigmine | Sugammadex
Started | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neostigmine | Sugammadex | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.16 (13.2) | 54.4 (13.5) | 53.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 15 | 14 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 28 | 28 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Incentive Spirometry Volume [Median (Inter-Quartile Range); unit: mL] | 2500 [2100 to 3500] | 2650 [2250 to 3500] | 2500 [2150 to 3500]
Hand Grip Strength [Mean (Standard Deviation); unit: psi] | 77.11 (27.8) | 74.4 (27.6) | 75.8 (27.5)
Preoperative ability to sit up [Count of Participants; unit: Participants] | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Incentive Spirometry, Change From Baseline and Recovery Profile - 30 Minutes
Description: Incentive spirometry measurements will be done at 30, 60 and 120 minutes after surgery. The change from baseline and recovery profile will be measured.
Time Frame: 30 Minutes
Population: The discrepancy between the number of participants analyzed and participate flow module is because patients were unable to perform this measure at this time point either due to significant sedation or significant pain
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Neostigmine | Sugammadex
Number analyzed (Participants) | 21 | 18
mL | -700 [-1650 to -250] | -862 [-1800 to -500]

2. Primary Outcome: Incentive Spirometry, Change From Baseline and Recovery Profile - 60 Minutes
Description: as for outcome 1
Time Frame: 60 Minutes after reversal
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Neostigmine | Sugammadex
Number analyzed (Participants) | 25 | 29
mL | -500 [-1300 to -250] | -1150 [-1850 to -362.5]

3. Primary Outcome: Incentive Spirometry, Change From Baseline and Recovery Profile - 120 Minutes
Description: as for outcome 1
Time Frame: 120 minutes after reversal
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Neostigmine | Sugammadex
Number analyzed (Participants) | 27 | 27
mL | -400 [-1560 to -200] | -850 [-1500 to -100]

4. Secondary Outcome: Grip Strength, Change From Baseline and Recovery Profile 30 Min
Description: Grip strength will be measured with a hand dynamometer
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: PSI
Arm/Group | Neostigmine | Sugammadex
Number analyzed (Participants) | 26 | 23
PSI | 24.15 (20.54) | 21.38 (20.0)

5. Secondary Outcome: Grip Strength, Change From Baseline and Recovery Profile 60 Min
Description: Grip strength will be measured with a hand dynamometer
Time Frame: 60 minutes after reversal
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: psi
Arm/Group | Neostigmine | Sugammadex
Number analyzed (Participants) | 28 | 29
psi | 12.68 (22.12) | 17.69 (15.76)

6. Secondary Outcome: Grip Strength, Change From Baseline and Recovery Profile 120 Min
Description: Grip strength will be measured with a hand dynamometer
Time Frame: 120 minutes after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: psi
Arm/Group | Neostigmine | Sugammadex
Number analyzed (Participants) | 28 | 29
psi | 7.84 (21.32) | 11.85 (14.53)

7. Secondary Outcome: Time to Extubation
Description: Measured time between surgery end and time of extubation (removal of breathing tube)
Time Frame: Immediately after surgery, up to 30 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Neostigmine | Sugammadex
Number analyzed (Participants) | 31 | 31
minutes | 8 [5 to 16] | 7 [4 to 11]

8. Secondary Outcome: Train of Four Ratio > 90% During PACU Admission
Description: Train of four ratio (TOFR) is the ration of the twitch height of the 4th twitch compared to the 1st twitch during train of four neuromuscular stimulation. This measurement was performed using a TOF Watch, which in an accelemyographer. Electric current is applied to the ulnar nevre and the twitches are measured in the thumb. Adequate reversal of neuromuscular blockade is defined as a TOFR >90%.
Time Frame: At PACU admission, approximately within one hour of reversal of neuromuscular blockade reversal.
Population: The discrepancy between the number of participants analyzed and participate flow module is because we were unable to obtain TOFR data for these patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Neostigmine | Sugammadex
Number analyzed (Participants) | 29 | 28
Participants | 25 | 25

9. Secondary Outcome: Quality of Recovery 15 Survey
Description: 15 question survey to assess patient's overall quality of recovery after anesthesia/surgery.
  Quality of Recovery 15 Survey. Minimum: 0 Maximum: 150 Higher Scores mean a better outcome and better quality of recovery.
  Part A: How have you been feeling in the last 24 hours? 0 = none of the time (poor), 10 = all of the time (excellent). Examples: able to breath easily, able to enjoy food, feeling rested. etc.
  Part B: Have you had any of the following in the last 24 hours? 10 to 0, where 10 = none of the time (Excellent) and 0 = all of the time (poor). Examples: moderate pain, nausea or vomiting, feeling worried or anxious, etc.
Time Frame: Postoperative day number one
Population: The discrepancy between the number of participants analyzed and participate flow module is because patients were unable to reach these patients on postoperative day number one.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Neostigmine | Sugammadex
Number analyzed (Participants) | 15 | 15
scores on a scale | 117 [99 to 128] | 105 [94 to 124]

10. Secondary Outcome: Time to Readiness for Post Anesthesia Care Unit (PACU) Discharge (Aldrete Score >9)
Description: Measured time between PACU admission and meeting PACU discharge readiness. PACU discharge was defined as when the patient had an Aldrete score of 9 or higher as determined by the PACU nurse. The Aldrete score is a measure of post anesthesia recovery. 0 is poor condition and 10 is excellent condition. There are 5 assessment items (able to move voluntary, breathing, consciousness, circulation (BP) and spO2) which are graded on a 0-2 point scale with 0 being poor and 2 being excellent.
Time Frame: Within 4 hours from the end of surgery
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Neostigmine | Sugammadex
Number analyzed (Participants) | 31 | 31
minutes | 109 [75 to 156] | 112 [77 to 158]

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Neostigmine | Sugammadex
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 2/31 | 2/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neostigmine (N=31) | Sugammadex (N=31)
Fever (General disorders) | 0 (0) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT02909439/Prot_SAP_000.pdf
  • Informed Consent Form (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT02909439/ICF_001.pdf